CLINICAL TRIAL: NCT04862845
Title: Effect of Combination of Duloxetine and Pregabalin to Improve Pain After Liposuction Surgery
Brief Title: Combination of Duloxetine and Pregabalin to Improve Postoperative Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor of anesthesia, SICU & and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: N-39-2021
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride; Pregabalin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients in group I (PD group) (Active Comparator)
  Interventions: Drug: Duloxetine and Pregabalin
- patients in group II (P group) (Active Comparator)
  Interventions: Drug: pregabalin
- patients in group III (C groups) (Sham Comparator)
  Interventions: Drug: sham

INTERVENTIONS:
Drug: Duloxetine and Pregabalin — will be received pregabalin with duloxetine 90 minutes preoperatively, then pregabalin every 12 hours with duloxetine once daily postoperatively until the fifth postoperative day.
  Arms: Patients in group I (PD group)
Drug: pregabalin — received pregabalin with a placebo capsule at 90 minutes preoperatively, then every 12 hours postoperatively with a placebo capsule once daily until the fifth postoperative day.
  Arms: patients in group II (P group)
Drug: sham — received two placebo capsules at 90 minutes preoperatively then placebo capsules every 12 hours, with one capsule daily postoperatively until the fifth postoperative day.
  Arms: patients in group III (C groups)

SUMMARY:
Postoperative pain is mediated by different mechanisms at multiple neural sites. Thus, multimodal analgesics can reduce the postoperative pain. Although Opioids are considered the analgesics of choice to treat moderate to severe pain, their use carries the risk of side effects and hyperalgesia. Multimodal analgesia can be achieved by combining different analgesics and different methods of administration, to provide better analgesia synergistically compared with conventional analgesia. Therefore,lower doses for each drug can be provided with fewer overall side-effects obtained from individual compounds.

Recently, antidepressants such as duloxetine, a selective serotonin and norepinephrine reuptake inhibitor (SSNRI), have accomplished pain relief in persistent and chronic pain as in fibromyalgia, postherpetic neuralgia, diabetic neuropathy, osteoarthritis and musculoskeletal pain. The analgesic effect of duloxetine is attributed to its ability to enhance both serotonin and norepinephrine neurotransmission in descending inhibitory pain pathways. Moreover, some studies have promoted its use to improve the quality of recovery after surgery and reduce the acute postoperative pain after knee replacement surgery , mastectomy , hysterectomy , and after spine surgery. In addition it can improve postoperative quality of recovery through mood improvement that can be helpful in the postoperative period.

The main objective of the present study was to examine perioperativelythe analgesic efficacy with the combination of duloxetine and prgabalinon postoperative pain when given as part of a multimodal pain strategy in patients undergoing surgery on liosuction. In addition to evaluating the patient's satisfaction and the adverse effects related to the combination of both medications.

ELIGIBILITY:
Inclusion criteria:

* Patients aged from 18 to40 years.
* ASA I-II.
* undergoing elective mega -liposuction surgery
* BMI from 18 to 50 kg/m2

  2. Exclusion criteria:
* Patient refusal
* Contraindication or chronic use (consistent use for longer than 3 months) to any of the study drugs ASA III-IV.
* Patients aged less than 18 or more than 50.
* Body mass index >50.
* Suffered from severe psychiatric disease or drug addiction;
* Chronic opioid consumption,
* a history of regular sedatives or anticonvulsants intake, serious organ disease or dysfunction
* inability to use a PCA device
* History of parenteral or oral analgesic intake within the last 48hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
total morphine consumption by ( mg ) | 72 hours
  intraoperative and initial 72 postoperative hours morphine consumption mg

SECONDARY OUTCOMES:
time to 1st request of rescue analgesia. | 24 hours
  Time to 1st request of rescue analgesia.
Postoperative pain score | 24 hous
  visual analog scale (VAS) score of pain (0 being 'no pain' and '10' being the maximal worst pain )
Postoperative Sedation Score | 24 hous
  postoperative sedation score assessed by the Modified Ramsay Sedation Score
Patient satisfaction | 72 hours
  Patient satisfaction 4-point scale (1 = poor, 2 = fair, 3 = good, 4 = excellent).
intraoperative and postoperative complication complications | 72 hours
  such as coughing, sedation, anxiety, ataxia, blurred vision, diplopia, nausea and vomiting, shivering, and dizziness was also recorded
Quality of Recovery questionnaire | 72 hours
  to assess preoperative health status

CONTACTS AND LOCATIONS:
Locations (1):
- facility of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided